CLINICAL TRIAL: NCT06501482
Title: "Interest of Postoperative Reintroduction of Chemotherapy in Patients Undergoing Resection of Colorectal Liver Metastases After Good Response to FOLFIRI-based Chemotherapy With or Without Targeted Agent" (Intergroup FRENCH- PRODIGE)
Brief Title: Adjuvant FOLFIRI Based-chemotherapy After Resection of CLM Responding to Preoperative FOLFIRI
Acronym: IRIMAD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220917; 2023-504831-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-27; First posted 2024-07-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Colorectal Liver Metastases
Keywords: Resected colorectal liver metastases; Response to preoperative chemotherapy; Postoperative FOLFIRI based chemotherapy; Disease-free survival
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: National, multicenter, open-label randomized, 2-arm, phase III superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative FOLFIRI group (Experimental): Irinotecan 180 mg/m2 + leucovorin 400 mg/m2 at day 1 then 5-FU 400 mg/m2 bolus followed by 2400 mg/m2 continuous infusion over 46 h biweekly. For a total of 12 cycles of perioperative chemotherapy including the preoperative chemotherapy
  Interventions: Drug: Postoperative reintroduction of FOLFIRI based chemotherapy
- No treatment group (control group) (No Intervention): No treatment

INTERVENTIONS:
Drug: Postoperative reintroduction of FOLFIRI based chemotherapy — Postoperative reintroduction of FOLFIRI: irinotecan 180 mg/m2 + leucovorin 400 mg/m2 at day 1 then 5-FU 400 mg/m2 bolus followed by 2400 mg/m2 continuous infusion over 46 h biweekly. For a total of 12 cycles of perioperative chemotherapy including the preoperative chemotherapy
  Arms: Postoperative FOLFIRI group

SUMMARY:
Eligible patients are patients with contraindication to preoperative oxaliplatin based-chemotherapy who underwent resection of no more than 10 colorectal liver metastases after preoperative FOLFIRI based chemotherapy with or without targeted agents. These patients must have objective response to treatment (radiologic or pathologic response). The standard care for these patients is no postoperative treatment although benefit of reintroduction of FOLFIRI chemotherapy in good responders could be expected.

This study is a National, multicenter, open-label randomized, 2-arm, phase III superiority trial comparing postoperative reintroduction of FOLFIRI based-chemotherapy (experimental arm) vs no treatment (control arm) in patients undergoing resection of colorectal liver metastases after good response to FOLFIRI-based chemotherapy with or without targeted agent.

The primary endpoint of the study is 3-year disease free survival. Based on published data, 3-year DFS in control group (absence of postoperative treatment is 25%. Expected 3-year DFS in the experimental group is 40%. The study will randomize 254 patients (127 in the chemotherapy group and 127 in the no treatment group) in 30 french academic centers.

DETAILED DESCRIPTION:
This study is a National, multicenter, open-label randomized, 2-arm, phase III superiority trial comparing postoperative reintroduction of FOLFIRI based-chemotherapy (experimental arm) vs no treatment (control arm) in patients undergoing resection of colorectal liver metastases after good response to FOLFIRI-based chemotherapy with or without targeted agent.

Inclusion criteria are:

* Histologically proven resected metachronous CLM with curative intent that could not be treated with perioperative oxaliplatin-based chemotherapy for oncologic or tolerability reasons. For this study, metachronous CLM is defined as liver recurrence occurring more than 12 months after treatment of the primary colorectal cancer.
* No more than 10 treated CLM at surgery
* At least 2 cycles and no more than 8 cycles of preoperative FOLFIRI based chemotherapy ± targeted therapy.
* Preoperative FOLFIRI based chemotherapy ± targeted therapy administered no more than 12 weeks before surgery
* R0/R1resection ± radiofrequency ablation with curative intent of all liver deposits with no macroscopic residual liver disease
* Objective response to preoperative therapy defined as complete or partial radiological response and/or major or complete pathologic response
* No extrahepatic or residual liver disease on baseline work-up including thoraco-abdominal CT scan within 6 weeks after surgery. 1 non-specific lung nodule of less than 10 mm in maximum diameter is not considered as extra-hepatic metastases
* Primary tumor (or liver metastasis) of CRC must be characterized for RAS and BRAF status
* No contraindication to FOLFIRI based chemotherapy
* Patients must be 18 years old or older
* A WHO performance status of 0 or 1
* Participants must be affiliated to a social security scheme The primary objective is demonstrate an improvement of disease-free survival rate at 3 years.

In the experimental arm, patients will be treated with irinotecan 180 mg/m2 + leucovorin 400 mg/m2 at day 1 then 5-FU 400 mg/m2 bolus followed by 2400 mg/m2 continuous infusion over 46 h biweekly. For a total of 12 cycles of perioperative chemotherapy including the preoperative chemotherapy.

In the control arm, patients do not receive any adjuvant treatment. This is an intention-to-treat trial. Based on published data, 3-year DFS in the control arm is 25%. Expected 3-year DFS in the experimental group is 40%. The sample size in each group is 127, with a total number of 185 events required, an exponential maximum likelihood test of equality of survival curves with a 0,050 two-sided significance level will have 80% power to detect the difference between groups (constant hazard-ratio of 0,662); assuming a 36 month length of accrual period, a 72 maximum length of follow up and 5% annual attrition (following exponential model) over study period (following exponential model) over study period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven resected metachronous CLM with curative intent that could not be treated with perioperative oxaliplatin-based chemotherapy for oncologic or tolerability reasons. For this study, metachronous CLM is defined as liver recurrence occurring more than 12 months after treatment of the primary colorectal cancer.
* No more than 10 treated CLM at surgery
* At least 2 cycles and no more than 8 cycles of preoperative FOLFIRI based chemotherapy ± targeted therapy.
* Preoperative FOLFIRI based chemotherapy ± targeted therapy administered no more than 12 weeks before surgery
* R0/R1resection ± radiofrequency ablation with curative intent of all liver deposits with no macroscopic residual liver disease
* Objective response to preoperative therapy defined as complete or partial radiological response and/or major or complete pathologic response
* No extrahepatic or residual liver disease on baseline work-up including thoraco-abdominal CT scan within 6 weeks after surgery. 1 non-specific lung nodule of less than 10 mm in maximum diameter is not considered as extra-hepatic metastases
* Primary tumor (or liver metastasis) of CRC must be characterized for RAS and BRAF status
* No contraindication to FOLFIRI based chemotherapy
* Patients must be 18 years old or older
* A WHO performance status of 0 or 1
* Participants must be affiliated to a social security scheme

Exclusion Criteria:

* Palliative/R2 resection of CLM
* 10 lesions or more treated at the time of surgery
* Patients undergoing only radiofrequency ablation of all liver deposit (this situation precludes the assessment of pathologic response to preoperative chemotherapy)
* Extra-hepatic or residual metastasis of CRC
* Absence of objective response to therapy (radiological or pathological response )
* Inflammatory bowel disease
* Known UGT1A1*28 allele homozygosity
* complete absence of dihydropyrimidine dehydrogenase (DPD) activity (blood uracil level ≥ 150 ng/ml
* Contraindications to investigational medicinal products (irinotecan, 5-FU, folinic acid) and to auxiliary medicinal products (ondansetron, methylprednisolone)
* Persistent toxicity ≥ grade 1 related to preoperative FOLFIRI based chemotherapy
* Known pregnancy (pregnancy test for women of childbearing) or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2028-06-27 (Estimated); Study Completion 2031-06-27 (Estimated)

PRIMARY OUTCOMES:
The disease-free survival rate | 3 years
  Disease-free survival rate at 3 years defined as the proportion of surviving patients without disease recurrence measured by Kaplan-Meier in the two treatment arms from the time to randomization. Disease-free survival will be defined as follows: time between randomization and disease recurrence or death whichever occurs first.
  In this trial, the disease-free survival is defined as the time to occurrence of first recurrence or death whatever comes first.
  Diagnosis of recurrence can be made only when the clinical and laboratory findings meet at least one of the criteria defined below:
  * Objective radiological recurrence on radiological imaging (ultrasound, CT scan, MRI scan, TEP scan as indicated by the clinical picture)
  * Positive cytology or biopsy (in case of ascites, anastomotic recurrence, doubt on radiological imaging) Note: an isolated elevated tumor marker level will not be considered acceptable evidence of cancer recurrence.
  * Death.

SECONDARY OUTCOMES:
The overall survival rate | 3 years
  All patients will be followed-up for at least 3 year after randomization or until death. Overall survival is defined as survival duration from the time of randomization to death. Patients who are still alive when last traced will be censored at the date of last follow-up.
The Liver-free survival rate | 3 years
  Liver-free survival is defined as survival duration from the time of randomization to first liver recurrence.

OTHER OUTCOMES:
The Extra -hepatic recurrence rate | 3 years
  The extra-hepatic recurrence rate is the rate of cancer relapse aside the liver. This rate will be evaluated at 3 years and at the date of last follow-up.
The safety including chemotherapy associated toxicity assessed by International Common Terminology Criteria for Adverse Events (CTCAE) grading system | At each cycle of postoperative FOLFIRI chemotherapy administration for a total of 12 cycles perioperative (including the preoperative chemotherapy) and each cycle is 15 days, then every 3 months for 2 years and then every 6 months for 3 years
  All adverse events will be recorded in the electronic case report form (eCRF) using the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 for adverse event reporting (see chapter 10. Safety assessment).
The compliance | At each cycle of postoperative FOLFIRI chemotherapy administration for a total of 12 cycles perioperative (including the preoperative chemotherapy) and each cycle is 15 days
  The ability to administrate a total of 12 cycles of FOLFIRI-based chemotherapy including preoperative treatment: Compliance with study protocol will be defined as completion of full dose planned preoperative treatment in each treatment arm. Any deviation and cause of deviation (toxicity, progression, physician or patient preference) from the protocol will be collected
The rate of treatment of recurrence | Every 3 months for 2 years and then every 6 months for 3 years
  Among patients who develop disease recurrence and who therefore achieved the primary endpoint, a proportion will be treated with curative intent including chemotherapy and local therapy (radiofrequency ablation or surgery). The proportion of patients undergoing treatment of recurrence with curative intent in will be evaluated in both groups
The quality of life | 1 year
  Quality of life assessed by QLQ C-30

CONTACTS AND LOCATIONS:
Overall Officials: Eric VICAUT, MHD, PHD, Study Chair — APHP; Eric VICAUT, MHD, PHD, Principal Investigator — APHP
Locations (1):
- Hôpital Kremlin Bicêtre, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No